CLINICAL TRIAL: NCT06891664
Title: Feasibility of Day-surgery Management for Patients Undergoing Robotic Radical Prostatectomy: a Randomized Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RS254/IRE/24
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day surgery management (Experimental): Day-surgery management of patients undergoing robotic radical prostatectomy. It represents a multidisciplinary management that includes nurses, physiotherapists, anesthesiologists and urologists. In addition, patients will be provided with a telemedicine device, to ensure contact between doctor and patient.
  Patients assigned to the experimental arm will be summoned together with the caregiver the days before the operation to discuss specifically with the nurse, anesthesiologist and urologist the procedure that they will have to follow. At this meeting, the functioning of the telemedicine device will be illustrated.
  Interventions: Procedure: Day surgery regimen for patients
- Ordinary management (Active Comparator): Management of patients undergoing robotic radical prostatectomy in an inpatient setting based on a minimum of two nights of hospitalization.
  Interventions: Other: Ordinary management

INTERVENTIONS:
Procedure: Day surgery regimen for patients — The protocol includes admission on the evening of Day -1 and the execution of the surgery on the morning of Day 0 under general anesthesia. The surgery will be performed with the aid of the Da Vinci Single-port robotic system with extraperitoneal access.
  Arms: Day surgery management
Other: Ordinary management — Management of patients undergoing robotic radical prostatectomy in an inpatient setting based on a minimum of two nights of hospitalization
  Arms: Ordinary management

SUMMARY:
To compare the day-surgery approach versus routine management in patients undergoing robotic radical prostatectomy, aimed at evaluating the feasibility of a one-day hospitalization regimen for robotic radical prostatectomy.

The study will allow to evaluate the patients'compliance and subsequently investigate the safety, the impact on the patient's quality of life and on the healthcare costs resulting from day-surgery management of patients undergoing robotic radical prostatectomy.

DETAILED DESCRIPTION:
The clinical study is aimed at evaluating the compliance of patients, candidates for robot-assisted radical prostatectomy for prostate cancer, to be enrolled in an RCT that provides for assignment to day surgery management (experimental arm) or ordinary management (control arm). The study involves the evaluation of the compliance of patients, candidates for robot-assisted radical prostatectomy for prostate cancer, to be enrolled in an RCT that provides for assignment to day surgery management (experimental arm) or ordinary management (control arm).

The study will allow us to test a protocol for day-surgery management that includes all the clinical and technological measures at our disposal, including single-port robotic surgery and telemedicine. Using the experience and results obtained from this trial, it will then be possible to design a confirmatory multicenter RCT that compares day-surgery management vs ordinary management. The latter will then have the task of demonstrating with a high level of evidence that robotic radical prostatectomy can be performed safely in day-surgery, guaranteeing economic advantages to the facility while also favoring a more rapid recovery of the patient. Considering that approximately 20,000 radical prostatectomies are performed every year in Italy, this paradigm shift could guarantee a significant economic advantage. A transition of this type requires robust scientific evidence in order to convince doctors, patients and health systems to rely on a more efficient health model based on better management of resources.

ELIGIBILITY:
Inclusion Criteria:

* patients with localized prostate adenocarcinoma at low-intermediate risk (EAU Risk classification);
* patients aged >= 18 years;
* patients with an indication to undergo robotic radical prostatectomy without lymphadenectomy according to the EAU guidelines;
* patients who agree to undergo robotic radical prostatectomy without lymphadenectomy according to the EAU guidelines by signing a written informed consent;
* patients eligible for robotic radical prostatectomy without lymphadenectomy and in the absence of contraindications to undergo the procedure;
* patient's ability to understand and willingness to sign a written informed consent indicating that he has understood the purpose and methods of conducting the study and is interested in participating.;
* patients able to follow the indications specified in the study protocol;
* patients domiciled (even temporarily) < 150 km away from the institution where the procedure will be performed;
* patients domiciled (even temporarily) < 60 minutes by car from a reference Emergency and Acceptance Department (DEA).

Exclusion Criteria:

* patients > 75 years of age;
* ASA > 2;
* second simultaneous surgery;
* prostate volume > 80 cc estimated on preoperative imaging (transrectal ultrasound or magnetic resonance imaging);
* patients receiving anticoagulants or oral antiplatelet drugs;
* other concomitant tumors undergoing treatment;
* previous pelvic radiotherapy;
* previous surgery for benign prostatic hypertrophy;
* patients lacking the digital literacy required to take advantage of telemedicine intervention;
* patients who cannot benefit from at least one caregiver;
* patients not suitable for a day-surgery approach based on the clinical evaluation of the operating surgeons and anesthetists.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-05-23 (Estimated); Study Completion 2027-05-23 (Estimated)

PRIMARY OUTCOMES:
Study enrollment rate among eligible patients. | 30 months
  RCT (randomized controlled trial) enrollment measured as the relative frequency percentage of patients who meet the eligibility criteria and agree to participate in the proposed trial (numerator), divided by the number of all eligible patients in the recruitment period (denominator). Patients who withdraw consent before knowing the outcome of randomization will be counted as having refused participation. The expected result is an enrollment rate of at least 30%. Therefore, the primary objective will be considered achieved if at least 30% of eligible patients agree to participate in the aforementioned trial

SECONDARY OUTCOMES:
Study Retention Rate | 30 months
  The retention rate will be measured as the relative percentage frequency of patients who remain in the study (numerator) of the total number of randomized patients (denominator). Patients who withdrew consent before knowing the outcome of randomization will be excluded from the denominator. In addition, the specific reasons for failure to remain will be listed. The retention rate will be compared between the two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Costantino Leonardo, Doctor, Principal Investigator — IRCCS National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy